CLINICAL TRIAL: NCT04642638
Title: Phase 2/3 Randomized, Blinded, Placebo-Controlled Trial to Evaluate the Safety, Immunogenicity, and Efficacy of INO-4800, a Prophylactic Vaccine Against COVID-19 Disease, Administered Intradermally Followed by Electroporation in Adults at High Risk of SARS-CoV-2 Exposure
Brief Title: Safety, Immunogenicity, and Efficacy of INO-4800 for COVID-19 in Adults at High Risk of SARS-CoV-2 Exposure
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated to prioritize Inovio's COVID-19 efforts to advance a heterologous booster strategy and optimize potential impact on global public health.
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: Advaccine (Suzhou) Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVID19-311; INNOVATE (Other: Inovio INO-4800 Vaccine Trial for Efficacy); WHO UTN: U1111-1266-9952 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-11-23; First posted 2020-11-24 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Coronavirus Infection; Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); COVID-19 Disease
Keywords: DNA vaccine; Electroporation; Healthy; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — reluscovtogene ralaplasmid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Phase 2: INO-4800 Dose Group 1 (Experimental): Participants received one ID injection of 1.0 milligram (mg) of INO-4800 followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Phase 2: INO-4800 Dose Group 2 (Experimental): Participants received two ID injections of 1.0 mg (total 2.0 mg per dosing visit) of INO-4800 followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Phase 2: Placebo Dose Group 1 (Placebo Comparator): Participants received one ID injection of placebo followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
  Interventions: Drug: Placebo; Device: CELLECTRA® 2000
- Phase 2: Placebo Dose Group 2 (Placebo Comparator): Participants received 2 ID injections of placebo followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
  Interventions: Drug: Placebo; Device: CELLECTRA® 2000
- Phase 3: INO-4800 Dose Group (2.0mg per dosing visit) (Experimental): Participants received two 1.0 mg ID injections of INO-4800, each followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Phase 3: Placebo Dose Group (Placebo Comparator): Participants received 2 ID injections of placebo per dosing visit, each followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
  Interventions: Drug: Placebo; Device: CELLECTRA® 2000

INTERVENTIONS:
Drug: INO-4800 — INO-4800 was administered ID on Day 0 and Day 28.
  Arms: Phase 2: INO-4800 Dose Group 1; Phase 2: INO-4800 Dose Group 2; Phase 3: INO-4800 Dose Group (2.0mg per dosing visit)
Device: CELLECTRA® 2000 — EP using the CELLECTRA® 2000 device was administered following ID delivery of INO-4800 on Day 0 and Day 28.
  Arms: Phase 2: INO-4800 Dose Group 1; Phase 2: INO-4800 Dose Group 2; Phase 3: INO-4800 Dose Group (2.0mg per dosing visit)
Drug: Placebo — Sterile saline sodium citrate (SSC) buffer (SSC-0001) was administered ID on Day 0 and Day 28.
  Other Names: SSC-0001; Placebo for INO-4800
  Arms: Phase 2: Placebo Dose Group 1; Phase 2: Placebo Dose Group 2; Phase 3: Placebo Dose Group
Device: CELLECTRA® 2000 — EP using the CELLECTRA® 2000 device was administered following ID delivery of sterile saline sodium citrate (SSC) buffer (SSC-0001) on Day 0 and Day 28.
  Arms: Phase 2: Placebo Dose Group 1; Phase 2: Placebo Dose Group 2; Phase 3: Placebo Dose Group

SUMMARY:
This is a Phase 2/3, randomized, placebo-controlled, multi-center trial to evaluate the safety, immunogenicity and efficacy of INO-4800 administered by intradermal (ID) injection followed by electroporation (EP) using CELLECTRA® 2000 device to prevent coronavirus disease 2019 (COVID-19) in participants at high risk of exposure to severe acute respiratory syndrome coronavirus - 2 (SARS-CoV-2).

The Phase 2 segment will evaluate immunogenicity and safety in approximately 400 participants at two dose levels across three age groups. Safety and immunogenicity information from the Phase 2 segment will be used to determine the dose level for the Phase 3 efficacy segment of the study involving approximately 7116 participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Working or residing in an environment with high risk of exposure to SARS-CoV-2 for whom exposure may be relatively prolonged or for whom personal protective equipment (PPE) may be inconsistently used, especially in confined settings.
* Phase 2 only: Screening laboratory results within normal limits for testing laboratory or are deemed not clinically significant by the Investigator.
* Be post-menopausal or be surgically sterile or have a partner who is sterile or use medically effective contraception with a failure rate of < 1% per year when used consistently and correctly from Screening until 3 months following last dose (Phase 2) or until last dose (Phase 3).

Key Exclusion Criteria:

* Acute febrile illness with temperature higher than or equal to 100.4°F (38.0°C) or acute onset of upper or lower respiratory tract symptoms (e.g., cough, shortness of breath, sore throat).
* Positive serologic or molecular (Reverse transcription polymerase chain reaction (RT-PCR)) test for SARS-CoV-2 at Screening (this criterion applies to all Phase 2 participants and only applies after approximately 402 participants positive for SARS-CoV-2 serologic test are randomized in the Phase 3 segment of the study).
* Pregnant or breastfeeding or intending to become pregnant or intending to father children within the projected duration of the trial starting from the Screening visit until 3 months following the last dose (Phase 2) or until last dose (Phase 3).
* Known history of uncontrolled human immunodeficiency virus (HIV) based on clusters of differentiation (CD4) count less than 200 cells per cubic millimeter (/mm^3) or a detectable viral load within the past 3 months.
* Is currently participating or has participated in a study with an investigational product within 30 days preceding Day 0.
* Previous or planned receipt of an investigational (including Emergency Use Authorization (EUA) or local equivalent authorization) or licensed vaccine for prevention or treatment of COVID-19, middle east respiratory syndrome (MERS), or severe acute respiratory syndrome (SARS) (documented receipt of placebo in previous trial would be permissible for trial eligibility).
* Respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease) requiring significant changes in therapy or hospitalization for worsening disease during the 6 weeks prior to enrolment.
* Immunosuppression as a result of underlying illness or treatment.
* Lack of acceptable sites available for ID injection and EP.
* Blood donation or transfusion within 1 month prior to Day 0.
* Reported alcohol or substance abuse or dependence, or illicit drug use (excluding marijuana use).
* Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Suaya, Study Director — Inovio Pharmaceuticals
Locations (27):
- United States (16):
  - Synexus Clinical Research US, Inc - Phoenix Southeast, Chandler, Arizona
  - Central Phoenix Synexus Clinical Research, Phoenix, Arizona
  - AMR Tempe, Tempe, Arizona
  - Optimal Research, LLC, San Diego, California
  - AMR South Florida, Coral Gables, Florida
  - Clinical Research Trials of Florida, Inc, Tampa, Florida
  - AMR Lexington, Lexington, Kentucky
  - Walter Reed Army Institute of Research, Silver Spring, Maryland
  - Ascension St. John Hospital, Detroit, Michigan
  - AMR Kansas City, Kansas City, Missouri
  - AMR, Clinical Research Consortium- Las Vegas, Las Vegas, Nevada
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tekton Research, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Advanced Clinical Research, West Jordan, Utah
- Colombia (5):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla, Atlántico
  - Clinica de la Costa LTDA, Barranquilla, Atlántico
  - Corazon IPS S.A.S, Barranquilla, Atlántico
  - Ips Centro Cientifico Asistencial Sas, Barranquilla, Atlántico
  - Centro de Investigaciones Clinicas IPS Cardiomet Pereira, Pereira, Risaralda Department
- Mexico (6):
  - BRCR Global Mexico, Guadalajara, Jalisco
  - Eukarya Pharmasite SC, Monterrey, Nuevo León
  - Unidad de Medicina Especializada SMA, San Juan del Río, Querétaro
  - Clinstile, SA de CV, Mexico City
  - SMIQ, S. de R. L. de C.V., Querétaro
  - FAICIC S. de R.L. de C.V., Veracruz

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 10 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the phase 2 segment, participants were enrolled at 16 study sites in the United States. For the Phase 3 segment, participants were enrolled at 11 study sites in Colombia and Mexico. They were enrolled between 30 November 2020 to 13 September 2022
Pre-assignment Details: In the Phase 2 segment, 618 participants were screened, of which 401 participants were enrolled to receive INO-4800 or placebo. In the Phase 3 segment, 978 participants were screened, of which 906 participants were enrolled to receive INO-4800 or placebo.
Groups:
- Phase 2: INO-4800 Dose Group 1: Participants received one intradermal (ID) injection of 1.0 milligram (mg) of INO-4800 followed by electroporation (EP) using the CELLECTRA® 2000 device on Day 0 and Day 28.
- Phase 2: INO-4800 Dose Group 2: Participants received 2 ID injections of 1.0 mg (total 2.0 mg per dosing visit) of INO-4800 followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
Period: Overall Study
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Started | 151 | 149 | 50 | 51 | 603 | 303
Intention-to-treat (ITT) Population (ITT population included all participants who were randomized.) | 151 | 149 | 50 | 51 | 603 | 303
Per Protocol (PP) Population (PP population included all participants who received all doses of the trial intervention and had no key protocol violations.) | 141 | 130 | 47 | 48 | 507 | 261
Safety Population (Safety population included all participants who received at least 1 dose of the trial intervention.) | 151 | 147 | 50 | 51 | 601 | 302
Completed | 110 | 98 | 35 | 39 | 0 | 0
Not Completed | 41 | 51 | 15 | 12 | 603 | 303
Not completed — Withdrawal by Subject | 23 | 29 | 9 | 7 | 61 | 27
Not completed — Lost to Follow-up | 17 | 18 | 5 | 5 | 6 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 10 | 3
Not completed — Reason Not Specified | 1 | 4 | 0 | 0 | 38 | 16
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Study Terminated | 0 | 0 | 0 | 0 | 484 | 250
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who were randomized.
Groups:
- Phase 2: INO-4800 Dose Group 1: Participants received one ID injection of 1.0 mg of INO-4800 followed by electroporation (EP) using the CELLECTRA® 2000 device on Day 0 and Day 28.
- Total: Total of all reporting groups
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group | Total
Number analyzed (Participants) | 151 | 149 | 50 | 51 | 603 | 303 | 1307
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-50 years | 98 | 97 | 32 | 34 | 533 | 267 | 1061
  Age: 51-64 years | 41 | 40 | 14 | 13 | 63 | 29 | 200
  Age: >=65 years | 12 | 12 | 4 | 4 | 7 | 7 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 77 | 28 | 30 | 245 | 120 | 576
  Male | 75 | 72 | 22 | 21 | 358 | 183 | 731
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 14 | 7 | 9 | 601 | 300 | 960
  Not Hispanic or Latino | 122 | 134 | 43 | 42 | 1 | 3 | 345
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 2 | 314 | 171 | 491
  Asian | 3 | 8 | 0 | 3 | 0 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 15 | 16 | 5 | 2 | 2 | 2 | 42
  White | 127 | 121 | 45 | 44 | 20 | 7 | 364
  More than one race | 2 | 2 | 0 | 0 | 267 | 123 | 394
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Change From Baseline in Antigen-specific Cellular Immune Response Measured by Interferon-gamma (IFN-γ) Enzyme-linked Immunospot (ELISpot) Assay
Description: Whole blood and serum samples were collected for the cellular immunology assessment. The antigen-specific cellular immune response to INO-4800 was measured in spot-forming units per million peripheral blood mononuclear cells (SFU/10^6, PBMC) using ELISpot. No samples collected after Week 6 were analyzed.
Time Frame: Baseline up to Week 6
Population: PP population included all participants who received all doses of the trial intervention and had no key protocol violations. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' denotes the number of participants available at individual timepoints.
Measure: Median (Full Range); unit: SFU/10^6, PBMC
Groups:
- Phase 2: INO-4800 Dose Group 1: Participants received one ID injection of 1.0 mg of INO-4800 followed by EP using the CELLECTRA® 2000 device on Day 0 and Day 28.
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2
Number analyzed (Participants) | 103 | 97 | 37 | 35
SFU/10^6, PBMC
  Baseline | 0.00 [0.0 to 90.0] | 2.20 [0.0 to 115.6] | 0.00 [0.0 to 25.6] | 0.00 [0.0 to 95.6]
  Change From Baseline at Week 6: number analyzed (Participants) | 96 | 91 | 35 | 31
  Change From Baseline at Week 6 | 6.70 [0.0 to 245.6] | 13.30 [0.0 to 311.1] | 0.00 [0.0 to 81.1] | 0.00 [0.0 to 54.4]
Statistical Analysis 1: Comparison: Phase 2: INO-4800 Dose Group 1 vs Phase 2: Placebo Dose Group 1; Test type: Other; Difference in median = 6.70, 95% CI 2-sided [0.00 to 6.70], Standard Error of Mean 3.35 — Post-baseline change from baseline in IFN-gamma ELISpot response magnitudes was compared between groups using differences in medians and associated non-parametric 95% confidence interval (CI)
Statistical Analysis 2: Comparison: Phase 2: INO-4800 Dose Group 2 vs Phase 2: Placebo Dose Group 2; Test type: Other; Difference in median = 13.30, 95% CI 2-sided [3.30 to 17.80], Standard Error of Mean 10.55 — Post-baseline change from baseline in IFN-gamma ELISpot response magnitudes was compared between groups using differences in medians and associated non-parametric 95% CI
Statistical Analysis 3: Comparison: Phase 2: INO-4800 Dose Group 1 vs Phase 2: INO-4800 Dose Group 2; Test type: Other; Difference in median = -6.60, 95% CI 2-sided [-10.00 to 0.00], Standard Error of Mean -5.00 — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Phase 2: Change From Baseline in Neutralizing Antibody Response Measured by a Pseudovirus-based Neutralization Assay
Description: The immune responses to INO-4800 were measured using assays that included a pseudovirus-based neutralization assay. Immunology blood samples were collected at serial timepoints. No samples collected after Week 6 were analyzed.
Time Frame: Baseline up to Week 6
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: inhibition dilution 50 (ID50)
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2
Number analyzed (Participants) | 133 | 120 | 47 | 45
inhibition dilution 50 (ID50)
  Baseline | 34.8 (0.42) | 40.6 (0.52) | 30.2 (0.40) | 38.0 (0.45)
  Change From Baseline at Week 6: number analyzed (Participants) | 133 | 119 | 47 | 45
  Change From Baseline at Week 6 | 3.1 (0.49) | 4.6 (0.52) | 1.2 (0.39) | 1.2 (0.49)
Statistical Analysis 1: Comparison: Phase 2: INO-4800 Dose Group 1 vs Phase 2: Placebo Dose Group 1; Test type: Other; Geometric Mean Fold Rise (GMFR) Ratio = 2.50, 95% CI 2-sided [1.720 to 3.632] — 95% CI of GMFR ratio is based on t-distribution, where GMFR ratio is based on the between-treatment-group comparisons
Statistical Analysis 2: Comparison: Phase 2: INO-4800 Dose Group 2 vs Phase 2: Placebo Dose Group 2; Test type: Other; GMFR Ratio = 3.88, 95% CI 2-sided [2.638 to 5.700] — 95% CI of GMFR ratio is based on t-distribution, where GMFR ratio is based on the between-treatment-group comparisons
Statistical Analysis 3: Comparison: Phase 2: Placebo Dose Group 1 vs Phase 2: Placebo Dose Group 2; Test type: Other; GMFR Ratio = 0.68, 95% CI 2-sided [0.512 to 0.893] — 95% CI of GMFR ratio is based on t-distribution, where GMFR ratio is based on the between-treatment-group comparisons

3. Primary Outcome: Phase 3: Percentage of Participants (SARS-CoV-2 Seronegative at Baseline) With Virologically-confirmed COVID-19 Disease
Description: Participants were virologically-confirmed cases of COVID-19, if tested positive by SARS-CoV-2 RT-PCR assay, with symptoms like fever (temperature of 100.4ºF/38.0ºC or higher), chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea, vomiting, diarrhoea. Participants with no prior exposure to COVID-19 at baseline were considered for the analysis.
Time Frame: From 14 days after completion of the 2-dose regimen up to 3 months post-dose 2 (i.e. Day 42 up to Day 126)
Population: For the Phase 3 segment, as pre-specified in the protocol, an independent endpoint adjudication committee (EAC) was to review and confirm the suspected COVID-19 cases which fulfilled the definition for virologically-confirmed COVID-19 cases. As the trial was prematurely terminated, suspected COVID-19 cases were not reconciled with the EAC. Therefore, data that was planned for the EAC to reconcile was not available for efficacy analysis and data could not be reported for the outcome measure.
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 2 and 3: Percentage of Participants With Solicited Injection Site Reactions
Description: Reactions arising from the injectable product administration procedure were reported as injection site reactions. Injection site reactions were assessed in accordance with the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials' (Food and Drug Administration [FDA] Guidance for Industry, September 2007). Participants were provided a diary to record the solicited injection site reactions. Local reactions to the injectable product such as pain, tenderness, erythema/redness, and induration/swelling were recorded. Injection site reactions were evaluated starting 30 minutes following the injection. The solicited injection site reactions were recorded for 7 days after each dose.
Time Frame: 7 days following each dose: Day 0 (Days 0 to Day 7) and Day 28 (Days 28 to Day 35)
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 151 | 147 | 50 | 51 | 601 | 302
percentage of participants
  Injection Site Pain | 27.2 | 36.1 | 20.0 | 23.5 | 19.1 | 21.2
  Injection Site Tenderness | 1.9 | 5.4 | 2.0 | 3.9 | 0 | 0
  Injection Site Erythema | 17.9 | 25.2 | 18.0 | 7.8 | 6.8 | 6.0
  Injection Site Swelling | 11.3 | 16.3 | 2.0 | 2.0 | 4.2 | 2.6

5. Secondary Outcome: Phase 2 and 3: Percentage of Participants With Unsolicited Injection Site Reactions
Description: Reactions arising from the injectable product administration procedure were reported as injection site reactions. Injection site reactions were assessed in accordance with the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials' FDA Guidance for Industry, September 2007. Local reactions to the injectable product such as pain, tenderness, erythema/redness, and induration/swelling were reported. Injection site reactions were evaluated starting 30 minutes following the injection. Unsolicited injection site reactions were recorded for up to 28 days after administration of dose 2.
Time Frame: From first dose of study drug up to Day 56
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 151 | 147 | 50 | 51 | 601 | 302
percentage of participants
  Injection Site Pain | 27.2 | 36.7 | 22.0 | 23.5 | 19.3 | 21.5
  Injection Site Tenderness | 0.6 | 0 | 0 | 1.9 | 0 | 0
  Injection Site Erythema | 17.9 | 25.2 | 18.0 | 7.8 | 6.8 | 6.0
  Injection Site Swelling | 11.3 | 16.3 | 2.0 | 2.0 | 4.2 | 2.6

6. Secondary Outcome: Phase 2 and 3: Percentage of Participants With Solicited Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a trial intervention that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Participants were provided a diary to record the solicited systemic AEs. The solicited AEs were recorded for 7 days after each dose.
Time Frame: 7 days following each dose: Day 0 (Days 0 to Day 7) and Day 28 (Days 28 to Day 35)
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 151 | 147 | 50 | 51 | 601 | 302
percentage of participants | 72.2 | 83.7 | 70.0 | 56.9 | 31.6 | 31.5

7. Secondary Outcome: Phase 2 and 3: Percentage of Participants With Unsolicited AEs
Description: An AE is defined as any untoward medical occurrence in a participant administered a trial intervention that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AEs were recorded for up to 28 days after administration of dose 2.
Time Frame: From first dose of study drug up to Day 56
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 151 | 147 | 50 | 51 | 601 | 302
percentage of participants | 74.2 | 85.0 | 74.0 | 62.7 | 38.8 | 37.1

8. Secondary Outcome: Phase 2 and 3: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a trial intervention that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or results in congenital anomaly or birth defect.
Time Frame: Phase 2: From first dose of study drug up to Day 393; Phase 3: From first dose of study drug up to Day 126
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 151 | 147 | 50 | 51 | 601 | 302
percentage of participants | 2.6 | 1.4 | 6.0 | 3.9 | 0.7 | 1.3

9. Secondary Outcome: Phase 2 and 3: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a trial intervention that does not necessarily have a causal relationship with this treatment. An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate.
Time Frame: Phase 2: From first dose of study drug up to Day 393; Phase 3: From first dose of study drug up to Day 126
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 151 | 147 | 50 | 51 | 601 | 302
percentage of participants | 0 | 0 | 0 | 2.0 | 0.3 | 0

10. Secondary Outcome: Phase 3: Number of Participants With Death From All Causes
Time Frame: Baseline up to Day 126
Population: Safety population included all participants who received at least one dose of the trial intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 601 | 302
Participants | 2 | 2

11. Secondary Outcome: Phase 3: Percentage of Participants (SARS-CoV-2 Seronegative at Baseline) With Non-Severe COVID-19 Disease
Description: The efficacy of INO-4800 in the prevention of COVID-19 disease was evaluated according to the degrees of COVID-19 disease severity in participants. Participants were confirmed cases of COVID-19, if tested positive by SARS-CoV-2 RT-PCR assay, with symptoms like fever (temperature of 100.4ºF/38.0ºC or higher), chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea, vomiting, diarrhoea. The case definition of severe COVID-19 was participants with COVID-19 having clinical signs at rest indicative of severe systemic illness, respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to an intensive care unit, or death. The case definition for non-severe COVID-19 was participants with confirmed COVID-19, and which did not meet the case definition of severe COVID-19.
Time Frame: From 14 days after completion of the 2-dose regimen up to 3 months post-dose 2 (i.e. Day 42 up to Day 126)
Population: For the Phase 3 segment, as pre-specified in the protocol, an independent EAC was to review and confirm the suspected COVID-19 cases which fulfilled the definition for virologically-confirmed COVID-19 cases. As the trial was prematurely terminated, suspected COVID-19 cases were not reconciled with the EAC. Therefore, data that was planned for the EAC to reconcile was not available for efficacy analysis and data could not be reported for the outcome measure.
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase 3: Percentage of Participants (SARS-CoV-2 Seronegative at Baseline) With Severe COVID-19 Disease
Description: The efficacy of INO-4800 in the prevention of COVID-19 disease was evaluated according to the degrees of COVID-19 disease severity in participants. Participants were confirmed cases of COVID-19, if tested positive by SARS-CoV-2 RT-PCR assay, with symptoms like fever (temperature of 100.4ºF/38.0ºC or higher), chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea, vomiting, diarrhoea. The case definition of severe COVID-19 was participants with COVID-19 having clinical signs at rest indicative of severe systemic illness, respiratory failure, evidence of shock, significant acute renal, hepatic, or neurologic dysfunction, admission to an intensive care unit, or death.
Time Frame: From 14 days after completion of the 2-dose regimen up to 3 months post-dose 2 (i.e. Day 42 up to Day 126)
Population: as for outcome 11
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase 3: Percentage of Participants (SARS-CoV-2 Seronegative at Baseline) With Death From COVID-19 Disease
Time Frame: From 14 days after completion of the 2-dose regimen up to 3 months post-dose 2 (i.e. Day 42 up to Day 126)
Population: as for outcome 11
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Phase 3: Percentage of Participants (SARS-CoV-2 Seropositive at Baseline) With Virologically-Confirmed SARS-CoV-2 COVID-19 Disease
Description: Participants were virologically-confirmed cases of COVID-19, if tested positive by SARS-CoV-2 RT-PCR assay, with symptoms like fever (temperature of 100.4ºF/38.0ºC or higher), chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea, vomiting, diarrhoea. Participants with prior exposure to COVID-19 at baseline were considered for the analysis.
Time Frame: From 14 days after completion of the 2-dose regimen up to 3 months post-dose 2 (i.e. Day 42 up to Day 126)
Population: as for outcome 11
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Phase 3: Change From Baseline in Antigen-specific Cellular Immune Response Measured by IFN-gamma ELISpot Assay
Description: Whole blood and serum samples were collected for the cellular immunology assessment. The antigen-specific cellular immune response to INO-4800 were measured using ELISpot.
Time Frame: Baseline up to Day 126
Population: Due to the early termination of the study, immunogenicity analysis that was pre-specified in the protocol was not performed in the Phase 3 segment of the study. Hence, data for this outcome measure was not collected.
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Phase 3: Change From Baseline in Neutralizing Antibody Response Measured by a Pseudovirus-based Neutralization Assay
Description: The immune responses to INO-4800 were measured using assays that included a pseudovirus-based neutralization assay.
Time Frame: Baseline up to Day 126
Population: as for outcome 15
Arm/Group | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Phase 2: From the first dose of the study drug up to Day 393; Phase 3: From the first dose of the study drug up to Day 126
Description: Safety population included all participants who received at least one dose of the trial intervention.
Arm/Group | Phase 2: INO-4800 Dose Group 1 | Phase 2: INO-4800 Dose Group 2 | Phase 2: Placebo Dose Group 1 | Phase 2: Placebo Dose Group 2 | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) | Phase 3: Placebo Dose Group
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/147 | 1/50 | 0/51 | 2/601 | 2/302
Serious Adverse Events (participants affected / at risk) | 4/151 | 2/147 | 3/50 | 2/51 | 4/601 | 4/302
Other Adverse Events (participants affected / at risk) | 115/151 | 127/147 | 42/50 | 38/51 | 279/601 | 140/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: INO-4800 Dose Group 1 (N=151) | Phase 2: INO-4800 Dose Group 2 (N=147) | Phase 2: Placebo Dose Group 1 (N=50) | Phase 2: Placebo Dose Group 2 (N=51) | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) (N=601) | Phase 3: Placebo Dose Group (N=302)
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 3
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: INO-4800 Dose Group 1 (N=151) | Phase 2: INO-4800 Dose Group 2 (N=147) | Phase 2: Placebo Dose Group 1 (N=50) | Phase 2: Placebo Dose Group 2 (N=51) | Phase 3: INO-4800 Dose Group (2.0mg Per Dosing Visit) (N=601) | Phase 3: Placebo Dose Group (N=302)
Injection site pruritus (General disorders) | 56 | 81 | 13 | 11 | 60 | 26
Injection site pain (General disorders) | 42 | 54 | 11 | 12 | 117 | 65
Fatigue (General disorders) | 44 | 57 | 22 | 11 | 0 | 0
Injection site erythema (General disorders) | 28 | 37 | 9 | 4 | 43 | 19
Injection site swelling (General disorders) | 17 | 24 | 1 | 1 | 0 | 0
Injection site bruising (General disorders) | 4 | 11 | 0 | 2 | 0 | 0
Chills (General disorders) | 6 | 3 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 6 | 3 | 0 | 33 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 49 | 13 | 9 | 39 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 28 | 5 | 4 | 0 | 0
Headache (Nervous system disorders) | 42 | 56 | 21 | 15 | 61 | 35
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 4 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 3 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 5 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 15 | 5 | 5 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 50 | 27
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 58 | 31
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 37 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT04642638/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT04642638/SAP_001.pdf